CLINICAL TRIAL: NCT03340675
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study With an Open-Label Extension to Determine the Safety, Pharmacokinetics and Efficacy of Oral Ifetroban in Subjects With Duchenne Muscular Dystrophy
Brief Title: Oral Ifetroban in Subjects With Duchenne Muscular Dystrophy
Acronym: DMD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-IFE-007; FD-R-6371 (Other Grant/Funding Number: FDA Orphan Products Development)
Record Dates: First submitted 2017-11-03; First posted 2017-11-13 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy Cardiomyopathy; Cardiomyopathy, Dilated
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — ifetroban

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind, dose-ranging
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each individual bottle is labelled with a unique numeric code that identifies the contents to the unblinded sponsor representative.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oral Ifetroban - Low Dose (Experimental): Weight based, once daily oral ifetroban
  Interventions: Drug: Ifetroban
- Oral Ifetroban - High Dose (Experimental): Weight based, once daily oral ifetroban
  Interventions: Drug: Ifetroban
- Placebos (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ifetroban — Weight based, once daily oral ifetroban
  Arms: Oral Ifetroban - High Dose; Oral Ifetroban - Low Dose
Drug: Placebo — Matching oral placebo
  Arms: Placebos

SUMMARY:
Duchenne muscular dystrophy (DMD) is a devastating X-linked disease which leads to loss of ambulation between ages 7 and 13, respiratory failure and cardiomyopathy (CM) at any age, and inevitably premature death of affected young men in their late twenties. DMD is the most common fatal genetic disorder diagnosed in childhood. It affects approximately 1 in every 3,500 live male births across all races and cultures, and results in 20,000 new cases each year worldwide.Significant advances in respiratory care have unmasked CM as the leading cause of death. As there are yet no specific cardiac treatments to extend life, the current study aims to address this unmet medical need using a new therapeutic strategy for patients with DMD.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
This is a phase 2 randomized, double-blind, placebo-controlled, multiple dose study with an optional open-label extension to determine the safety, pharmacokinetics (PK) and efficacy of two doses of oral ifetroban in subjects with DMD. DMD patients who meet the inclusion criteria and none of the exclusion criteria will receive oral ifetroban or placebo once daily for 12 months. Subjects will be enrolled into one of three treatment groups, low-dose ifetroban, high-dose ifetroban or placebo. Each dose level will be evaluated by eight subjects with early stage (LVEF > 45%) DMD-associated cardiomyopathy and eight subjects with more advanced stage (LVEF 35-45%) cardiac disease as there may be differences in the treatment effect based on cardiac involvement. Each subject treated will be evaluated for first-dose and steady-state exposure PK. All subjects who receive treatment will be assessed for safety. All subjects with at least one efficacy assessment post-baseline will be evaluated for efficacy. Blood and urine will be collected for standard and novel cardiac biomarkers. Target enrollment met for early-stage subjects (LVEF > 45%); study closed to enrollment prior to meeting target enrollment in the late-stage cohort (LVEF 35-45%). All subjects who complete the 12-month study are eligible to enter an optional open label extension period consisting of treatment with high-dose ifetroban only. Subjects in the open label extension will be evaluated for safety and cardiac efficacy every 12 months.

ELIGIBILITY:
Inclusion criteria:

1. Males 7 years of age and older with the diagnosis of DMD, defined as phenotype consistent with DMD and either positive genotype, first degree relative with positive genotype, or confirmatory muscle biopsy.
2. Stable dose of oral corticosteroids for at least 8 weeks or has not received corticosteroids for at least 30 days.
3. Stable cardiac function defined as change in left ventricular ejection fraction (LVEF) of < 15% and no heart failure admission over the last 12 months; LVEF 35% or greater by cine cardiac magnetic resonance imaging (MRI) or echocardiography; myocardial damage in one or more left ventricular segments evident by late gadolinium enhancement allowed; concurrent angiotensin-converting enzyme inhibitors (ACEI), beta-blocker (BB) or angiotensin receptor blocker (ARB) therapy allowed (selection of which dictated by clinical care) if started three months or greater from first dose of IMP without change in dose. Aldosterone receptor antagonists (eg. Spironolactone or eplerenone) allowed if started 12 months or greater from first dose of Investigational Medicinal Product (IMP). No changes throughout the study allowed, except in the event of a decline in left ventricular ejection fraction (LVEF) >5% following the baseline CMR as measured by a subsequent CMR at the same center. Should this occur, changes in cardiac medications are allowed on the study.

   a. Late-stage cohort: Subjects are eligible for the late-stage cohort if the subject has: i. LVEF 35%-45% by cine cardiac magnetic resonance imaging (MRI) or echocardiography or ii. historically documented LVEF 35%-45% by cine cardiac magnetic resonance imaging (MRI) or echocardiography and if their baseline MRI is less than 50%.
4. Subjects aged 18 years and older, informed consent obtained directly. For subjects ages 7-17 years old (yo), both assent from the subject and permission from a parent or guardian.

Exclusion criteria:

1. Clinically significant illness other than DMD
2. Clinically significant laboratory abnormality not associated with DMD
3. Major surgery within six weeks prior to the first dose of study drug, or planned surgery during this study which would interfere with the ability to perform study procedures
4. Require antiarrhythmic therapy and/or initiation of diuretic therapy for management of acute heart failure in the last 6 months
5. A LVEF of < 35% by Cardiac Magnetic Resonance Imaging (CMR) and/or fractional shortening of < 15% based on echocardiography (ECHO) during screening
6. A known bleeding disorder or has received anticoagulant treatment within 2 weeks of study entry
7. Allergy to gadolinium contrast or known renal insufficiency defined as abnormal cystatin C or creatinine above the upper limit of normal for age. The male serum reference ranges as follows:

   * Age 7-9 years - 0.2-0.6 mg/dL
   * Age 10-11 years - 0.3-0.7 mg/dL
   * Age 12-13 years - 0.4-0.8 mg/dL
   * Age 14-15 years - 0.5-0.9 mg/dL
   * Age 16 years or older - 0.8-1.3 mg/dL
8. Non-MR compatible implants (e.g. neurostimulator, automatic implantable cardioverter-defibrillator [AICD])
9. Subjects who participated in a therapeutic clinical trial within 30 days or five half-lives (whichever is longer) of study entry
10. Any other condition that could interfere with the subject's participation

Min Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Markham, MD, Principal Investigator — Riley Children's Hospital
Locations (10):
- United States (10):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Mattel Children's Hospital, Los Angeles, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Saint. Louis Children's Hospital, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Monroe Carrell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitchell R, Frederick NE, Holzman ER, Agobe F, Allaway HCM, Bagher P. Ifetroban reduces coronary artery dysfunction in a mouse model of Duchenne muscular dystrophy. Am J Physiol Heart Circ Physiol. 2021 Jul 1;321(1):H52-H58. doi: 10.1152/ajpheart.00180.2021. Epub 2021 May 28. PMID 34048282

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized 1:1:1 to receive either high dose ifetroban, low dose ifetroban, or matching placebo daily for 52 weeks.
Pre-assignment Details: 46 participants were randomized into the study
Groups:
- High Dose Ifetroban: Oral ifetroban, 150 mg or 300 mg daily for 52 weeks (Subjects weighing < 35 kg received 150 mg or ≥ 35 kg received 300 mg ifetroban)
- Low Dose Ifetroban: Oral ifetroban, 50 mg or 100 mg daily for 52 weeks (Subjects weighing < 35 kg received 50 mg or ≥ 35 kg received 100 mg ifetroban)
- Placebo: Oral placebo daily for 52 weeks
Period: Double Blind
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
Started (Five participants were randomized into the study but withdrew prior to receiving treatment (No longer interested in study = 4; Withdrawn by site = 1)) | 18 (The relationship of IMP to adverse events leading to withdrawal were adjudicated to be 'Unlikely Related' or 'Unrelated' except for two participants in the High Dose Ifetroban group with events of 'Contusion' noted as 'Probably Related' and one participant in the Placebo group with an event of 'Headache' noted as 'Probably Related') | 12 | 11 (The relationship of IMP to adverse events leading to withdrawal were adjudicated to be 'Unlikely Related' or 'Unrelated' except for two participants in the High Dose Ifetroban group with events of 'Contusion' noted as 'Probably Related' and one participant in the Placebo group with an event of 'Headache' noted as 'Probably Related')
Completed | 13 | 9 | 8
Not Completed | 5 | 3 | 3
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Period: Open Label Extension
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
Started | 13 | 9 | 8
Completed | 10 | 7 | 8
Not Completed | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo | Total
Number analyzed (Participants) | 18 | 12 | 11 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.2 (5.9) | 17.3 (5.8) | 14.7 (4.9) | 17.0 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 18 | 12 | 11 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 16 | 12 | 10 | 38
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 4
  Not Hispanic or Latino | 17 | 12 | 8 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 54.3 (17.9) | 53.2 (20.7) | 42.4 (16.9) | 50.8 (18.8)
BMI (kg/m^2) [Count of Participants; unit: Participants]
  < 18.5 (Underweight) | 3 | 0 | 3 | 6
  18.5 - 24.9 (Normal weight) | 7 | 7 | 5 | 19
  25.0 - 29.9 (Overweight) | 5 | 3 | 1 | 9
  ≥ 30 (Obese) | 3 | 2 | 2 | 7
BMI Z-scores [Mean (Standard Deviation); unit: Z-score] — BMI Z-score indicating the number of standard deviations a participant's BMI is from the average BMI for their age and sex. A Z-score of 0 indicates the average BMI with positive Z-scores being above and negative Z-scores being below the mean. A Z-score > -2 or <2 is typically considered healthy.
  Z-score | 0.62 (1.4) | 1.1 (0.71) | 0.15 (2.2) | 0.59 (1.6)
Ambulatory [Count of Participants; unit: Participants]
  Yes | 8 | 4 | 4 | 16
  No | 10 | 8 | 7 | 25
Ventilatory Support [Count of Participants; unit: Participants]
  Yes | 2 | 2 | 0 | 4
  No | 16 | 10 | 11 | 37
Stage of DMD [Count of Participants; unit: Participants]
  Early (LVEF > 45%) | 14 | 11 | 11 | 36
  Late (LVEF 35 - 45%) | 4 | 1 | 0 | 5
Background DMD Therapy [Count of Participants; unit: Participants]
  No background therapy | 2 | 1 | 1 | 4
  Steroids only | 11 | 6 | 6 | 23
  ASO only | 0 | 0 | 0 | 0
  Steroids + ASO | 5 | 5 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: Percentage of subjects with one or more treatment emergent adverse event
Time Frame: Baseline through 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
Number analyzed (Participants) | 18 | 12 | 11
Participants
  Any TEAE | 14 | 9 | 10

2. Secondary Outcome: Pharmacokinetics Area Under the Curve
Description: Plasma ifetroban and its acyl glucuronide metabolite were measured pre-dose and at 0.5, 1.0, 4.0, 8.0 and 24.0 h post dose on Day 0 and pre-dose and 0.5 h post-dose on Day 7. Area under the curve until the last measurement was calculated for the plasma concentration versus time curves for ifetroban and its acyl glucuronide metabolite after administration of assigned oral ifetroban dose
Time Frame: Pre-dose and at 0.5, 1.0, 4.0, 8.0 and 24.0 h post-dose on Day 0 and pre-dose and 0.5 h post-dose on Day 7
Population: Fewer participants are represented here due to missing assessments for this measure.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban
Number analyzed (Participants) | 13 | 8
h*ng/mL
  Ifetroban | 3196 (2485) | 761 (585)
  Ifetroban Glucuronide | 45116 (30211) | 13789 (9700)

3. Secondary Outcome: Pharmacokinetics Maximum Serum Concentration (Cmax)
Description: Plasma ifetroban and its acyl glucuronide metabolite were measured pre-dose and at 0.5, 1.0, 4.0, 8.0 and 24.0 h post dose on Day 0 and pre-dose and 0.5 h post-dose on Day 7 to determine the maximum plasma concentration of ifetroban and its acyl glucuronide metabolite after administration of assigned oral ifetroban dose
Time Frame: Pre-dose and at 0.5, 1.0, 4.0, 8.0 and 24.0 h post dose on Day 0 and pre-dose and 0.5 h post-dose on Day 7
Population: Fewer participants are represented here due to missing assessments for this measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban
Number analyzed (Participants) | 13 | 8
ng/mL
  Ifetroban | 1560 (2028) | 272 (300)
  Ifetroban Glucuronide | 9787 (7148) | 2276 (1955)

4. Secondary Outcome: Pharmacokinetics Time to Reach Cmax (Tmax) Concentration
Description: Plasma ifetroban and its acyl glucuronide metabolite were measured pre-dose and at 0.5, 1.0, 4.0, 8.0 and 24.0 h post dose on Day 0 and pre-dose and 0.5 h post-dose on Day 7 to determine the time to maximum plasma concentration of ifetroban and its acyl glucuronide metabolite following administration of assigned oral ifetroban dose
Time Frame: Pre-dose and at 0.5, 1.0, 4.0, 8.0 and 24.0 h post dose on Day 0 and pre-dose and 0.5 h post-dose on Day 7
Population: Fewer participants are represented here due to missing assessments for this measure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban
Number analyzed (Participants) | 13 | 8
h
  Ifetroban | 0.71 (0.24) | 1.09 (1.2)
  Ifetroban Glucuronide | 2.81 (6.43) | 1.89 (2.47)

5. Secondary Outcome: Pharmacokinetics Plasma Terminal Half-life Concentration
Description: Plasma ifetroban were measured pre-dose and at 0.5, 1.0, 4.0, 8.0 and 24.0 h post dose on Day 0 and pre-dose and 0.5 h post-dose on Day 7. The terminal elimination half-life was calculated from the plasma concentration versus time curves for ifetroban following administration of assigned oral ifetroban dose
Time Frame: Pre-dose and at 0.5, 1.0, 4.0, 8.0 and 24.0 h post dose on Day 0 and pre-dose and 0.5 h post-dose on Day 7
Population: Fewer participants are represented here due to missing assessments for this measure.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban
Number analyzed (Participants) | 7 | 4
h | 12.96 (5.73) | 8.99 (4.6)

6. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction
Description: Change from baseline at month 12 in left ventricular ejection fraction
Time Frame: Baseline visit and Month 12 visit
Population: Differences in number of participants analyzed is due to missing evaluations at one or more timepoint
Measure: Mean (Standard Deviation); unit: Percentage of LVEF
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
Number analyzed (Participants) | 12 | 7 | 6
Percentage of LVEF | 1.8 (5.44) | 0 (5.16) | -1.5 (3.27)

7. Secondary Outcome: Change From Baseline in FEV1
Description: Change from baseline at month 12 in Forced Expiratory Volume in 1 second
Time Frame: Baseline through month 12
Population: Differences in number of participants analyzed is due to missing evaluations at one or more timepoint
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
Number analyzed (Participants) | 13 | 9 | 7
Liters | -0.05 (0.233) | -0.11 (0.294) | 0.01 (0.169)

8. Secondary Outcome: Change From Baseline in Percent Predicted FEV1
Description: Change from baseline at month 12 in percent predicted Forced Expiratory Volume in 1 second
Time Frame: Baseline through month 12
Population: Differences in number of participants analyzed is due to missing evaluations at one or more timepoint
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
Number analyzed (Participants) | 13 | 9 | 7
Percent | -1.92 (10.67) | -7.89 (9.226) | -3.29 (6.775)

9. Secondary Outcome: Change From Baseline in FVC
Description: Change from baseline at month 12 in Forced Vital Capacity
Time Frame: Baseline through month 12
Population: Differences in number of participants analyzed is due to missing evaluations at one or more timepoint
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
Number analyzed (Participants) | 13 | 9 | 7
Liters | -0.08 (0.291) | -0.07 (0.378) | -0.08 (0.291)

10. Secondary Outcome: Change From Baseline in Percent Predicted FVC
Description: Change from baseline at month 12 in percent predicted Forced Vital Capacity
Time Frame: Baseline through month 12
Population: Differences in number of participants analyzed is due to missing evaluations at one or more timepoint
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
Number analyzed (Participants) | 13 | 9 | 7
Percent | -3.31 (10.491) | -6.11 (11.050) | -8.14 (15.700)

11. Secondary Outcome: Change From Baseline in Maximal Expiratory Pressure
Description: Change from baseline at month 12 in maximal expiratory pressure
Time Frame: Baseline through month 12
Population: Differences in number of participants analyzed is due to missing evaluations at one or more timepoint
Measure: Mean (Standard Deviation); unit: cm of water
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
Number analyzed (Participants) | 13 | 8 | 6
cm of water | -1.69 (8.625) | 2.00 (16.466) | -16.50 (25.774)

12. Secondary Outcome: Change From Baseline in Maximal Inspiratory Pressure
Description: Change from baseline at month 12 in maximal inspiratory pressure
Time Frame: Baseline through month 12
Population: Differences in number of participants analyzed is due to missing evaluations at one or more timepoint
Measure: Mean (Standard Deviation); unit: cm of water
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
Number analyzed (Participants) | 13 | 8 | 6
cm of water | -6.00 (7.000) | -9.13 (8.935) | 1.17 (20.14)

13. Secondary Outcome: Change From Baseline in Peak Expiratory Flow Rate
Description: Change from baseline at month 12 in peak expiratory flow rate
Time Frame: Baseline through month 12
Population: Differences in number of participants analyzed is due to missing evaluations at one or more timepoint
Measure: Mean (Standard Deviation); unit: Liters/second
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
Number analyzed (Participants) | 13 | 6 | 6
Liters/second | 0.09 (0.643) | -0.19 (0.414) | 0.51 (0.844)

14. Secondary Outcome: Change From Baseline in Percent Predicted Peak Expiratory Flow Rate
Description: Change from baseline at month 12 in percent predicted peak expiratory flow rate
Time Frame: Baseline through month 12
Population: Differences in number of participants analyzed is due to missing evaluations at one or more timepoint
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
Number analyzed (Participants) | 12 | 6 | 5
Percent | -3.58 (15.395) | -3.83 (11.250) | 2.40 (20.477)

15. Secondary Outcome: Change From Baseline in Quality-of-life
Description: The Pediatric Quality of Life Inventory (PedQL) questionnaire measures core dimensions of health as delineated by the World Health Organization.
  The core module includes 23 items comprising 14 dimensions. The Gastrointestinal module includes 74 items comprising 14 dimensions. The Neuromuscular module includes 25 items comprising 3 dimensions. Each item in the modules is measured on a 5-point Likert scale of 0-4 with 0 indicating 'never' and 4 indicating 'almost always'.
  The Likert scores for each subscale are reversed scored and linearly transform to a 0-100 scale with 0=100, 1-75, 2=50, 5=25, and 4=0.
  A higher score indicates better health-related quality of life. Subscale scores are averaged to generate the total score reported with a range of 0-100.
  Results are presented as change from baseline at 12 months. The questionnaire was completed by the participant and the parent/guardian of the participant.
Time Frame: Baseline through 12 months
Population: Differences in number of participants analyzed is due to missing evaluations at one or more timepoint
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
Number analyzed (Participants) | 14 | 10 | 9
Scores on a scale
  Generic Core Module (Participant Response): number analyzed (Participants) | 14 | 8 | 7
  Generic Core Module (Participant Response) | -0.06 (15.9) | 4.39 (11.5) | -4.03 (13.1)
  Generic Core Module (Parent Response): number analyzed (Participants) | 12 | 8 | 7
  Generic Core Module (Parent Response) | -7.62 (14.3) | 0.43 (19.6) | -11.4 (21.5)
  Gastrointestinal Module (Participant Response): number analyzed (Participants) | 14 | 9 | 7
  Gastrointestinal Module (Participant Response) | -7.08 (22.7) | 4.08 (6.45) | -2.03 (10.7)
  Gastrointestinal Module (Parent Response): number analyzed (Participants) | 13 | 8 | 7
  Gastrointestinal Module (Parent Response) | 4.20 (6.59) | -0.03 (7.62) | -5.57 (4.95)
  Neuromuscular Module (Participant Response): number analyzed (Participants) | 14 | 9 | 7
  Neuromuscular Module (Participant Response) | 1.31 (10.4) | 3.49 (13.0) | 1.93 (12.0)
  Neuromuscular Module (Parent Response): number analyzed (Participants) | 13 | 8 | 7
  Neuromuscular Module (Parent Response) | 7.77 (8.01) | 2.00 (6.74) | -6.57 (10.3)

ADVERSE EVENTS:
Time Frame: From initiation of treatment through study completion, up to 1 year
Arm/Group | High Dose Ifetroban | Low Dose Ifetroban | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 3/18 | 2/12 | 2/11
Other Adverse Events (participants affected / at risk) | 14/18 | 9/12 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Ifetroban (N=18) | Low Dose Ifetroban (N=12) | Placebo (N=11)
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Ifetroban (N=18) | Low Dose Ifetroban (N=12) | Placebo (N=11)
Nausea (Gastrointestinal disorders) | 2 | 2 | 3
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 4 | 1 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 2
Pneumonia (Infections and infestations) | 2 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Muscle contracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 3
Dizziness (Nervous system disorders) | 2 | 0 | 0
Ejection fraction decreased (Investigations) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Delayed puberty (Endocrine disorders) | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT03340675/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT03340675/SAP_001.pdf